CLINICAL TRIAL: NCT03305640
Title: Identification of an Atypical acetabuLar frActure With an Independent Roof Component: Incidence and Description
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ALARIC
Record Dates: First submitted 2017-10-02; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: acetabular fracture surgery — acetabular fracture surgery

SUMMARY:
Treatment of acetabular fractures needs a perfect diagnosis to anticipate surgical difficulties. E. Letournel described a rare atypical both-column fracture which " introduces enormous surgical difficulties ". Its particularity is a sagittal comminution interesting the acetabular roof.

In this experience the particular fracture is probably under-diagnosed. The purpose of this study is to give the exact incidence and a precise description of these fractures to improve their surgical management.

ELIGIBILITY:
Inclusion Criteria:

* patient with acetabular fracture

Exclusion Criteria:

* other type of fracture

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: every patient with acute acetabular fractures managed in a single institution between 2007 and 2013
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
measurement of volume-rendered 3D-CT images on preoperative CT-scans | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pomme JOUFFROY, MD, Principal Investigator — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France